CLINICAL TRIAL: NCT00100360
Title: 5HT1A and SERT Imaging During Pharmacologically Induced Hypogonadotropic Hypogonadism With and Without Estrogen and Progesterone Replacement
Brief Title: Hormonal Causes of Menstrual-Related Mood Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050059; 05-M-0059
Record Dates: First submitted 2004-12-29; First posted 2004-12-30 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2016-12-15

CONDITIONS: Mood Disorders; Depression
Keywords: Gonadal Steroids; GnRH Agonist; Depression; Menstrual Cycle; Menstrually Related Mood Disorder; MRMD; Healthy Volunteer; HV
MeSH Terms: conditions — Mood Disorders; Depression

SUMMARY:
This study will explore possible hormonal causes of menstrual-related mood disorders (MRMD) by stopping the menstrual cycle with a drug called Lupron and then giving in sequence two menstrual cycle hormones, progesterone and estrogen. The study will first evaluate Lupron's effectiveness in treating MRMD and will then examine the effects of giving estrogen and progesterone on mood and behavior. In addition, positron emission tomography (PET) and magnetic resonance imaging (MRI) will be used to study serotonin receptors and transporters - molecules in the brain that are thought to play a major role in mood changes related to the menstrual cycle.

Menstruating women between 18 and 50 years of age who are in good health, not pregnant, and not taking medications may be eligible for this study. Women with MRMD must have had at least moderately severe MRMD or behavioral disturbances for at least 6 months within 2 years of entering the study. Healthy controls must have no history of MRMD or behavioral disturbances. Candidates undergo physical and neurological examinations, chest x-ray, electrocardiogram, and blood and urine tests. Results of a recent Pap smear (no longer than 12 months before beginning the study) must be available.

Participants undergo the following tests and procedures:

* Drug treatment: Lupron is injected into a muscle once a month for 5 months. After the second month, participants receive estrogen or progesterone, or both, daily. Estrogen is delivered through a skin patch (20 micrograms per day) and the progesterone is taken as a rectal or vaginal suppository twice a day for the remaining 12 weeks of the study. Every day, all participants wear a skin patch and insert two suppositories, but at some point during the 12 weeks, active medication is replaced with placebo to allow the drugs to wash out of the body.
* Physical examination and blood draw: A physical examination and blood tests are done at the start of the study and several times during the study to assess general health, evaluate liver and kidney function, and measure blood cell counts.
* Response to treatment drugs: Responses to Lupron, estrogen, and progesterone are evaluated periodically with interviews and symptoms self-rating scales. Control subjects also take paper and pencil psychological tests.
* PET imaging: A total of six PET scans are done at three time points during hormone treatment. PET uses small amounts of a radioactive chemical called a tracer that "labels" active areas of the brain. For the procedure, the subject lies on the scanner bed. A special mask is fitted to the head and attached to the bed to help keep the subject's head still during the scan so the images will be clear. A brief scan is done just before the radioactive tracer is injected to help in analyzing the PET data. After the tracer is injected through a catheter (plastic tube) placed in the arm, pictures are taken for about 2 hours, during which the subject lies still on the scanner bed.
* MRI scan: MRI uses a magnetic field and radio waves to produce images of body tissues and organs. For this procedure, the patient lies on a table that is moved into the scanner (a narrow cylinder) and wears earplugs to muffle loud knocking and thumping sounds that occur during the scanning process. The procedure lasts about 1 hour.

DETAILED DESCRIPTION:
The central serotonergic (5HT) system is one of the candidate systems that may mediate the abnormal mood and behavioral response to ovarian steroids observed in women with menstrual-related mood disorders (MRMD). Numerous studies have attempted to measure 5HT system function in women with MRMD and controls; however, previous studies were restricted to the evaluation of indirect measures of 5HT function (e.g., platelet 5HT uptake or responses to serotonergic pharmacologic challenges). Radioligand imaging of specific components of the 5HT system currently represents the most direct measure of central serotonergic function available. In this study we will image serotonergic measures during pharmacological conditions previously demonstrated to induce a remission and a subsequent provocation of mood symptoms in women with MRMD but not controls.

This protocol has two outcome measures (5HT(1A) binding and SERT binding), two groups of subjects (women with MRMD and controls), and three distinct hormonal conditions (hypogonadism, estrogen replacement, and progesterone replacement). Our principal aim in this study is to investigate differences in the outcome measures in women with MRMD compared to controls. Our primary hypothesis is that 5HT(1A) binding will be decreased and SERT binding will be increased in women with MRMD. A secondary hypothesis is that women with MRMD, but not controls, will display reproductive steroid modulation of 5HT(1A) and SERT binding. This study will help test existing hypotheses about the pathophysiologic relevance of serotonin function in MRMD and the role of reproductive steroids in serotonergic regulation. First, we selected 5HT(1A) receptor binding as an outcome measure for the following reasons: 5HT(1A) function is modulated by both estradiol and progesterone, abnormalities of 5HT(1A) binding have been reported in both depressive and anxiety disorders as well as possibly MRMD, 5HT(1A) receptors have been identified as potential mediators of estradiol's antidepressant-like effects in the forced swim test, and the 5HT(1A) system is involved in the regulation of GABA activity abnormalities of which have been implicated in MRMD. Second, we selected SERT binding as an outcome measure for the following reasons: selective serotonin reuptake inhibitors, but not traditional antidepressants, are effective treatments for MRMD; abnormalities of SERT binding have been reported in depressive disorders in women, preliminary data suggest that women with MRMD are characterized by an elevated frequency of the long, more transcriptionally active polymorphism of the serotonin transporter (5HTTLPR) (Roca et al); women with MRMD have altered imipramine binding and platelet 5HT uptake compared to controls as well as altered platelet paroxetine binding (which normalize with successful treatment with GnRH agonist); and, finally, SERT message, binding and protein have been reported to be changed by ovarian steroids in preclinical studies.

We hypothesize that the effects of hormonal condition on 5HT(1A) (receptor) binding will differ in patients and controls. Specifically, we anticipate that 5HT1A binding will be decreased in hippocampus and prefrontal cortex in patients with MRMD but not controls. Such a decrease, if a trait characteristic, will be demonstrable irrespective of hormonal state. However, as symptoms of MRMD are directly precipitated by estradiol or progesterone (see below), it is possible that symptoms are accompanied by state and steroid-dependent changes in 5HT(1A) binding and function. Consequently, our secondary hypothesis is that estradiol or progesterone induces changes in 5HT(1A) (receptor) binding in women with MRMD but not in control women.

Similarly, we hypothesize that women with MRMD will have increased SERT binding activity compared to controls, consistent with the therapeutic efficacy of selective serotonin reuptake inhibitors in this condition. However, a secondary hypothesis is that estradiol or progesterone-induced changes in SERT binding will occur in a hormone-dependent and mood state-dependent manner. Specifically, consistent with the literature in rodents, acute changes in ovarian steroids will increase SERT binding in association with the induction of symptoms in women with MRMD but not controls.

ELIGIBILITY:
* INCLUSION CRITERIA:

Women who meet the criteria for MRMD will have participated in Protocol No. 81-M-0126, The Evaluation of Women with Menstrually Regulated Mood and Behavior Disorders:

Women with MRMD:

* History within the last two years of at least six months with menstrually-related mood or behavioral disturbances of at least moderate severity-i.e., disturbances that are distinct in appearance and associated with a notable degree of subjective distress.
* Symptoms should have a sudden onset and offset.
* age 18-50.
* Not pregnant and in good medical health.
* Medication free.
* No prior DSM-IV Axis I disorder.
* No prior history of treatment with antidepressant medications

All patients participating in this protocol will have already participated in protocol No. 81-M-0126 and will have a prospectively confirmed and predictable relationship between their mood disorder and the premenstrual phase of the menstrual cycle; i.e., a 30% change in severity of symptom self rating scales, relative to the range of the scale employed, during the seven days premenstrually compared with the seven days post-menstrually in two out of three months of study.

Women without MRMD:

* No history of menstrual-related mood or behavioral disturbances;
* Age 18 and 50 years;
* Not pregnant;
* Good medical health;
* Medication free.
* The absence of menstrual-related mood disorders will be prospectively confirmed during a two month period prior to the study entry when subjects will complete daily visual analogue rating scales monitoring both mood and behavior as outlined in NIMH protocol # 81-M-0126.
* The Structured Clinical Interview for DSM-IV will be administered to all women prior to study entry. Any patient or control with a current and any control with a past Axis I psychiatric diagnosis will be excluded from participating in this protocol.
* Prior to treatment, a complete physical and neurological examination will have been performed (with normal chest X-ray and EKG) and the following routine laboratory data obtained:

A. Blood

--Complete blood count; thyroid function tests; renal function tests, such as BUN and creatinine; electrolytes; glucose; liver function tests, B-hCG for pregnancy test.

B. Urine

* Routine urinalysis.
* GnRH agonist will not be administered to any subject with significant clinical or laboratory abnormalities.
* Additional tests and exclusion criteria.
* Results of PAP smear performed not longer than 12 months prior to onset of treatment will be obtained. Subjects taking birth control pills or diuretics will be excluded from the study, as will patients taking psychotropic agents (e.g., lithium carbonate, tricyclic antidepressants). All subjects will be required to use non-hormonal forms of birth control (e.g., barrier methods) to avoid pregnancy during this study.

EXCLUSION CRITERIA:

The following conditions will constitute contraindications to treatment with hormonal therapy and will preclude a subject's participation in this protocol.

* History consistent with endometriosis.
* Diagnosis of ill-defined, obscure pelvic lesions, particularly undiagnosed ovarian enlargement.
* Hepatic disease as manifested by abnormal liver function test.
* History of mammary carcinoma.
* History of pulmonary embolism or phlebothrombosis.
* Undiagnosed vaginal bleeding.
* Porphyria.
* Diabetes mellitus.
* History of malignant melanoma.
* Cholecystitis or pancreatitis.
* Cardiovascular or renal disease.
* Pregnancy.
* Any woman meeting the Stages of Reproductive Aging Workshop Criteria (STRAW) for the perimenopause. Specifically, we will exclude any woman with an elevated plasma FSH level (> 14 IU/L) and with menstrual cycle variability of > 7 days different from their normal cycle length.

Further, subjects will be warned not to become pregnant during the study and will be required to employ barrier contraceptive methods.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2004-12-22; Study Completion 2016-12-15

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Schmidt, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] McEwen BS, Alves SE. Estrogen actions in the central nervous system. Endocr Rev. 1999 Jun;20(3):279-307. doi: 10.1210/edrv.20.3.0365. No abstract available. PMID 10368772
- [Background] Osterlund MK, Halldin C, Hurd YL. Effects of chronic 17beta-estradiol treatment on the serotonin 5-HT(1A) receptor mRNA and binding levels in the rat brain. Synapse. 2000 Jan;35(1):39-44. doi: 10.1002/(SICI)1098-2396(200001)35:13.0.CO;2-T. PMID 10579806
- [Background] Lu NZ, Bethea CL. Ovarian steroid regulation of 5-HT1A receptor binding and G protein activation in female monkeys. Neuropsychopharmacology. 2002 Jul;27(1):12-24. doi: 10.1016/S0893-133X(01)00423-7. PMID 12062903